CLINICAL TRIAL: NCT06722989
Title: The Impact of Mobile Application-guided Physical Exercise in Healthy Pregnant Women on Vital Physiological Parameters Measured with a Wearable Tracking Device
Brief Title: The Impact of Mobile Application-guided Physical Exercise on Physiological Parameters in Healthy Pregnant Women
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tanja Premru-Srsen, Assoc. Prof., University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 0120-47/2024-2711-6
Record Dates: First submitted 2024-11-15; First posted 2024-12-09 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Pregnancy
Keywords: pregnacy; physical activity; physical exercise; wearable tracking device; mobile guided exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mobile-guided exercise group (Experimental): Exercises for pregnant women in the SG will fall into moderate physical activity. They will be previously assessed by a perinatologist with a license to guide exercise during pregnancy. Each exercise will last 30 minutes, including initial warm-up exercises and final stretching exercises.
  The recommended moderate activity for pregnant women is at least 150 minutes per week, achieved on at least three days. For pregnant women aged 29 years or less, this means within the limits of a heart rate of 125 to 146 beats/min. For pregnant women aged 30 years or more, it is within the limits of a heart rate of between 121 and 141 beats per minute. According to the Borg scale of perceived exertion from six to 20, moderate exercise is rated between 13 and 14, corresponding to the specified heart rate thresholds. The pregnant woman will rate her exercise on the Borg perceived exertion scale from six to 20. The recommended number of steps per day will be at least 6,000.
  Interventions: Behavioral: mobile-guided exercise
- Unguided physical activity (Active Comparator): In this arm, pregnant women will be physically active at their discretion.
  Interventions: Behavioral: Unguided physical activity

INTERVENTIONS:
Behavioral: mobile-guided exercise — Exercises for pregnant women in the SG will fall into moderate physical activity. They will be previously assessed by a perinatologist with a license to guide exercise during pregnancy. Each exercise will last 30 minutes, including initial warm-up exercises and final stretching exercises.
  The recommended moderate activity for pregnant women is at least 150 minutes per week, achieved on at least three days. For pregnant women aged 29 years or less, this means within the limits of a heart rate of 125 to 146 beats/min. For pregnant women aged 30 years or more, it is within the limits of a heart rate of between 121 and 141 beats per minute. According to the Borg scale of perceived exertion from six to 20, moderate exercise is rated between 13 and 14, corresponding to the specified heart rate thresholds. The pregnant woman will rate her exercise on the Borg perceived exertion scale from six to 20. The recommended number of steps per day will be at least 6,000.
  Arms: mobile-guided exercise group
Behavioral: Unguided physical activity — In this group, pregnant women will be physically active at their discretion.
  Arms: Unguided physical activity

SUMMARY:
After the second-trimester anomaly scan, healthy pregnant women will be offered inclusion in the study. Before inclusion, participants will fill out a questionnaire on the suitability of moderate physical exercise. After signing the consent form for the study, they will receive a random wrist-tracking device. The investigators will inform them about the use and possibilities of the wrist-tracking device. Suppose they will be randomly assigned to the group with a guided exercise program for pregnant women. In that case, they will also have a guided exercise program via a mobile application, where they will receive one of the exercises intended for pregnant women every day for up to 30 minutes. The investigators will also present and explain all the exercises to them, emphasizing the crucial role they play in our study. The investigators will also explain when they should stop exercising and immediately consult a perinatologist on the phone number provided. If they are randomly assigned to the control group, they will not receive exercise, but they can be physically active at their discretion.

DETAILED DESCRIPTION:
The research will be a randomized intervention study on the impact of physical activity on physiological parameters and sleep duration during pregnancy. The research will be designed as a naturalistic study based on the guidelines for assessing the appropriateness of heart rate measurements with wrist-based heart rate monitors in biobehavioral research. The study will be conducted at the Gynecology Clinic at the University College of Medicine in Ljubljana.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years,
* confirmed duration of pregnancy with ultrasound measurement between the crown and the coccyx of the fetus in the first trimester,
* legal capacity,
* understanding of the Slovenian and English languages,
* signed consent form for the study, access to encrypted data, and use of data according to GDPR.

Exclusion Criteria:

pregnant women who will not sign a consent form for the study and the GDPR.

* pregnant women who will not allow the use of the key to access encrypted measurement data
* women under the influence of illegal substances (drugs or alcohol) that may interfere with their ability to participate and comply with the investigation procedures,
* any acute or chronic disease, disorder or condition, including cognitive dysfunction,
* pregnant women with multiple pregnancies,
* pregnant women with conditions that constitute a contraindication to regular physical exercise during pregnancy:

  * with a cervix < 30 mm,
  * with persistent unexplained bloody discharge,
  * with a placenta < 30 mm from the internal os,
  * with a growth-restricted fetus,
  * with rupture of the amniotic sac,
  * with a previous premature birth < 32 weeks,
  * with recurrent miscarriages
  * with one or more affirmative answers in the self-assessment questionnaire for physical fitness.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting heart rate variability | From enrolment to the end of treatment at 5 weeks.
  Heart rate variability (HRV) refers to the change in the interval between two beats (beat-to-beat interval) and allows a non-invasive assessment of the balance between the cardiac sympathetic and parasympathetic nervous systems. It will be measured during rest (sleep).

SECONDARY OUTCOMES:
Resting cardiac coherence | From enrolment to the end of treatment at 5 weeks.
  Cardiac coherence, or physiological coherence, describes a measure of the stability and harmony of individual oscillatory regulatory systems in the body at any given time. It is reflected in the regular, sine-wave pattern of the heartbeat. It will be measured during rest (sleep).
Resting heart rate | From enrolment to the end of treatment at 5 weeks.
  Heart rate measured during sleep.
Sleep duration | From enrolment to the end of treatment at 5 weeks.
  Overall duration of sleep and deep sleep duration.
Systemic vascular resistance (SVR) | At the enrolment and conclusion of the study after 5 weeks.
  Systemic vascular resistance is the quantitative value for left ventricular afterload. In most patients, changes in vascular resistance reflect changes in arteriolar tone or changes in the viscosity of blood. It will be measured by USCOM.
BMI z-score | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
AST/ALT ratio | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Fasting triglycerides | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Fasting glucose | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Fasting HDL | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Single-Point Insulin Sensitivity Estimator (SPISE) | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity
Quantitative Insulin Sensitivity Check Index (QUICKI) | At the enrolment and conclusion of the study after 5 weeks.
  Measure of Insulin sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Premru-Srsen, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- UMCLjubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared on request.
Supporting Information: Study Protocol
Time Frame: From study completion.
Access Criteria: Upon request and review of the request.